CLINICAL TRIAL: NCT05017259
Title: The Metabolomic Exploration of Low-carbohydrate and Calorie Restriction Diet on Weight Reduction, Post weigh-in Recovery and Exercise Performance in Taekwondo Athletes
Brief Title: Calorie Restriction Diets on Weight Reduction, Post weigh-in Recovery and Exercise Performance in Athletes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chin Hsu (Other)
Responsible Party: Sponsor-Investigator, Chin Hsu, Assistant professor, National Taiwan Sport University
Organization: National Taiwan Sport University (Other)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MOST 108-2410-H-028-005
Record Dates: First submitted 2021-08-15; First posted 2021-08-23 (Actual); Last update posted 2021-08-23 (Actual); Status verified 2021-08

CONDITIONS: Diet, Reducing
MeSH Terms: interventions — Caloric Restriction

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- low carbohydrate trial (Experimental): The energy distribution was carbohydrate 10%, protein 40-50%, fat 40-50% in the LC trial.
  Interventions: Dietary Supplement: calorie restriction diet
- high carbohydrate trial (Active Comparator): The energy distribution was carbohydrate 60-65%, protein 30-40%, fat 5-10% in the HC trial.
  Interventions: Dietary Supplement: calorie restriction diet

INTERVENTIONS:
Dietary Supplement: calorie restriction diet — The 7-day low-calorie diet contained 15.8 ± 0.4 kcal/kg/d in both trials, divided into three meals a day.

SUMMARY:
Low-carbohydrate diets are often used as weight-loss strategies by obese individuals and athletes. This diet has effects on oxidizing fat and suppressing appetite. But short term evidences are still few. In combat sports such as taekwondo, athletes prefer rapid weight loss to achieve a desired weight category. The purpose of this study was to investigate the impact of the low carbohydrate diet combined with strict calorie restriction on body composition and exercise performance in taekwondo athletes.

DETAILED DESCRIPTION:
This study used a randomized cross-over design. Each participant completed a low carbohydrate and a high carbohydrate trial in a random order, separated by a 30-day wash-out period. Each trial comprised of a 7-day weight loss period, followed by an 18-hr recovery period. The purpose of this study was to investigate the effect of 7-day caloric restriction with low- or high-carbohydrate diet, combined with an 18-hr recovery period, on body weight loss and taekwondo-specific performance.

ELIGIBILITY:
Inclusion Criteria:

* Must have at least 6 years of Taekwondo training experience
* Must have participated in domestic or international competitions

Exclusion Criteria:

* Smoking
* Cardiovascular disease
* Diabetes
* Hypertension
* Any medication in the past 3 months

Ages: 20 Years to 24 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2019-08-17 (Actual); Primary Completion 2019-09-26 (Actual); Study Completion 2019-09-26 (Actual)

PRIMARY OUTCOMES:
Body weight in kilograms assessed by air-displacement plethysmography (Bod Pod) | 1 min
  The body weight (kg) of participants was determined before and after calorie restriction intervention to evaluate the degree of weight loss.
Body fat mass in kilograms assessed by air-displacement plethysmography (Bod Pod) | 1 min
  The body fat mass (kg) of participants was determined before and after calorie restriction intervention to evaluate the degree of weight loss.
Lean body mass in kilograms assessed by air-displacement plethysmography (Bod Pod) | 1 min
  The lean body fat mass (kg) of participants was determined before and after calorie restriction intervention to evaluate the degree of weight loss.

SECONDARY OUTCOMES:
Taekwondo-specific reaction time in seconds assessed by Electromyography (EMG) signals | 1 min
  The reaction time (sec) was measured before and after weight loss to assess the difference in exercise performance. The participants were asked to make the fist on the left hand as soon as they see a light signal, then start the taekwondo-specific movement. The reaction time was calculated as the time from the beginning of the light signal to the start of electromyography (EMG) signal of the left thenar muscles. The movement was performed 5 times. The average reaction time was used to arrive at one reported value.

CONTACTS AND LOCATIONS:
Overall Officials: Chin Hsu, Principal Investigator — Assistant professor
Locations (1):
- National Taiwan University of Sport, Taichung, Taiwan

IPD SHARING:
Plan to Share IPD: No